CLINICAL TRIAL: NCT06654284
Title: Patient-Reported Quality of Life in Patients With an Implantable-Cardioverter Defibrillator - A Longitudinal Observational Study
Acronym: QoL-ICD II
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S69418
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Implantable Cardioverter Defibrillator (ICD)
Keywords: quality of life; Implantable Cardioverter Defibrillator (ICD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of life questionnaires — All patients will receive a combination of quality of life questionnaires aimed at predeifined time points (baseline, 3 months, 1 year, 3 year, 6 year, 9 year and 12 year) collecting a complete overview of different aspects of quality of life, including: - Florida patient acceptance score (FPAS) - Short Form Health Survey (SF-12) - Kansas City Cardiomyopathy Questionnaire (KCCQ-12) - Hospital Anxiety and Depression Scale (HADS) - Florida Shock Acceptance score (FSAS) - Steinke Sexual Concerns Inventory - the "Good Death" questionnaire

SUMMARY:
Patients at risk for life-threatening arrhythmias are eligible for the implantation of an implantable cardioverter-defibrillator (ICD), which has repeatedly shown improved survival. However, living with an ICD may pose several challenges and affect quality of life (QoL). This prospective longitudinal observational cohort studies will provide detailed insights in the change of patient-reported QoL after ICD impalntation. The aim is to study the change in time of the QoL perspective of patients who have an ICD, including physical and emotional health; ICD acceptance; concerns of ICD patients with regard to physical and sexual activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Patients either scheduled for a new ICD implantation or scheduled for an elective generator change
* Willing and able to provide signed written informed consent.

Exclusion Criteria:

* Patients with a mental disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any type of implantable cardioverter-defibrillator implanted and followed at UZ Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2042-12 (Estimated); Study Completion 2042-12 (Estimated)

PRIMARY OUTCOMES:
General QoL assessed using the Short Form Health Survey (SF-12) | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  General QoL assessed using the Short Form Health Survey (SF-12)
  The SF-12 measures the experienced health or health-related quality of life. The SF-12 is a shortened version of the longer SF-36. This questionnaire consists of twelve items, divided into eight subcategories:
  - General Health
  * Physical Functioning
  * Role Physical
  * Role Emotional
  * Bodily Pain
  * Mental Health
  * Vitality
  * Social functioning For each subcategory, a score between 0 and 100 is calculated using an available key. This score can then be compared to an available normative population. Average values below 50 indicate poorer physical/mental health compared to that normative population, while values above 50 indicate better health.

SECONDARY OUTCOMES:
- Cardiac-specific QoL assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  The KCCQ-12 is a shortened, but validated version of the KCCQ-23, and measures symptoms, physical and social limitations, and quality of life in patients with heart failure.2 The 12 questions have variable answer options, but all are based on a Likert scale. KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Florida Shock Acceptance score (FSAS) | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  Florida Shock Acceptance score (FSAS) The FSAS is intended to measure ICD shock anxiety.4 The measure was designed by an interdisciplinary team including electrophysiology and clinical psychology. Items were based on clinical experience with ICD patients. The scale itself consists of 10 items which respondents rate on a five-point Likert scale ranging from 1 (not at all) to 5 (all of the time). The score of the FSAS is determined by summing the items with higher values representing greater shock anxiety and lower values representing lower shock anxiety.
ICD acceptance assessed using the Florida Patient Acceptance Survey (FPAS) | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  The primary endpoint of the cross-sectional QoL-ICD study is the ICD acceptance assessed using the Florida Patient Acceptance Survey (FPAS). The FPAS began as a self-report survey with 47 items composed with the help of experts on psychosocial functioning in device patients, an expert in the field of psychometrics, and a cardiac electrophysiologist.2 Information obtained through surveys and interviews were used as guidelines for item construction. The result is an 18 question survey. Of these 18 questions, there are 3 filler items which are still relevant for ICD patients and the remaining questions cover 4 domains: (1) Return to Function; (2) Device-Related Distress; (3) Positive Appraisal; and (4) Body Image Concerns. Items are rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). Scale scores were calculated for each of the factors. By combining the scores for each question, a total FPAS score can be calculated.
Steinke Sexual Concerns Inventory | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  Steinke Sexual Concerns Inventory (SSCI, general cardiac version) The SSCI is an instrument that consists of 9 items reflecting change in the sexual relationship, sexual fears, change in sexual interest, symptoms associated with sexual activity, sexual dysfunction and any other sexual concerns.5 The items are rated on a scale of 0 to 3, where 0 indicates 'never' and 3 indicates 'frequently'. Higher scores indicate greater sexual concerns. Based on previous research, three potential subscales (sexual fears, symptoms, sexual dysfunction) were identified among the items.
"Concept of a Good Death" questionnaire | baseline, 3 months, 1 year, 3 years, 6 years, 9 years, adn 12 years
  The Concept of a Good Death measures three distinct domains, reflecting the psychosocial/spiritual, physical, and clinical aspects of a good death. The surveys comprises 17 questions on a 4-point Likert scale ranging from 'not at all' to 'essential'.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided